CLINICAL TRIAL: NCT03800771
Title: DOuble tasK Test On ergometeR - Basic Research on Acceptability and Use
Acronym: DOKTORBRAU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018-A01109-46
Record Dates: First submitted 2018-12-20; First posted 2019-01-11 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Elderly Patients
Keywords: geriatric; dual-task; ergometer

STUDY DESIGN:
Intervention Model Description: Patients are inhomogeneous in term of cognitive and physical function. The aim is to test faisability and security thus investigator will include a relatively large amount of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Practice dual-task tests (Experimental): The study consists to practice these dual-task tests with a new device which name is "Cycléo BRAU" that allows to the patients to achieve carefully an attentional task: cycle. Results will be compared tothe results obsvered during the routine GAITRITE analysis ( a validated tool for elderly patients and gait analysis).
  Interventions: Device: Cycléo BRAU; Device: GAITRITE®

INTERVENTIONS:
Device: Cycléo BRAU — Practice dual-task tests.
Device: GAITRITE® — Routine practice dual-task tests.

SUMMARY:
The goal of the study is to show the concordance between the dual-task test achieved usually on an electronic treadmill and the dual-task test achieved with a cyclo-ergometer.

DETAILED DESCRIPTION:
Usually, dual task tests are only achieved on electronic treadmills. Patients who are coming to perform these tests are mainly subjects with various levels of cognitive disorders and with a high risk of fall because of potential motor and cognitive disorders.

The investigator will select patients referred for double task walking tests. After the walking test, investigator will perform dual-task tests with a new bicycle device "Cycléo BRAU" which allows the patients to achieve mental tasks while cycling. The aim of using a bicycle is to limit the risk of falls compared to the treadmill or walking task. The "Cycléo BRAU" device is equiped with a video projector which projects an environment of virtual reality. It allows cycling without resistence and thus is not based on any incremental worload. The mental tasks on bicycle will be of increasing difficulty and parameters such as cycling speed will be recorded. Loss of speed regularity will be considered as an abnormal response. The task for which cycling is stopped will be recorded and compared to the results of the usual walking test.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years old
* Patient with a near visual acuity upper or equal to 2/10
* Patient with a score of MMSE upper than 10
* Patient able to walk on a treadmill for 15 meters on straight line without help
* Patient covered by the French health insurance
* Patient (or support person or legal representative) able to understand the protocol
* Patient (or support person or legal representative) agrees to be involve in the protocol and sign the consent form

Exclusion Criteria:

* Patient has a wash-out period for another clinical trial
* Patient with a medical contraindication to practice bicycle
* Patient with locomotor disorders preexisting, whatever the reason
* Patient needing extern help to walk like a walking frame, rollator or tricycle
* Patient with a medical or surgical disease acute from less of 3 months
* Patient with cerebrovascular accident history or any other cerebro-medullary diseases with sensorimotor consequences
* Patient with severe depression (Geriatric Depression Scale 15 items upper than 10)
* Patient with a low proficiency of French (oral or written)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2022-05-17 (Actual)

PRIMARY OUTCOMES:
Speed | 12 months
  Evaluate the concordance of the speed during the tests on treadmill and on cyclo-ergometer.
Speed variability | 12 months
  Evaluate the concordance the speed variability during the tests on treadmill and on cyclo-ergometer.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, MD; PhD, Principal Investigator — University Hospital in Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided